CLINICAL TRIAL: NCT01068964
Title: Safety and Efficacy of Bimatoprost Timolol Ophthalmic Solution in Patients With Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192024-052
Record Dates: First submitted 2010-02-12; First posted 2010-02-17 (Estimated); Results first posted 2012-01-20 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 0.03% Bimatoprost/0.5% Timolol in Same Bottle (Experimental): Bottle 1: 0.03% Bimatoprost/0.5% Timolol Ophthalmic Solution Bottle 2: Vehicle Ophthalmic Solution
  Interventions: Drug: 0.03% Bimatoprost/0.5% Timolol Ophthalmic Solution
- 0.03% Bimatoprost and 0.5% Timolol in Separate Bottles (Active Comparator): Bottle 1: 0.03% Bimatoprost Ophthalmic Solution Bottle 2: 0.5% Timolol Ophthalmic Solution
  Interventions: Drug: 0.03% Bimatoprost Ophthalmic Solution and 0.5% Timolol Ophthalmic Solution

INTERVENTIONS:
Drug: 0.03% Bimatoprost/0.5% Timolol Ophthalmic Solution — One drop from each bottle, administered once daily in the evening for 4 weeks Bottle 1: 0.03% Bimatoprost/0.5% Timolol Ophthalmic Solution Bottle 2: Vehicle Ophthalmic Solution
  Other Names: Bottle 1: Ganfort®
  Arms: 0.03% Bimatoprost/0.5% Timolol in Same Bottle
Drug: 0.03% Bimatoprost Ophthalmic Solution and 0.5% Timolol Ophthalmic Solution — One drop from each bottle, administered once daily in the evening for 4 weeks Bottle 1: 0.03% Bimatoprost Ophthalmic Solution Bottle 2: 0.5% Timolol Ophthalmic Solution
  Other Names: Bottle 1: Lumigan®; Bottle 2: Timoptol®
  Arms: 0.03% Bimatoprost and 0.5% Timolol in Separate Bottles

SUMMARY:
This study will evaluate the safety and efficacy of once daily administered 0.03% Bimatoprost/0.5% Timolol Ophthalmic Solution compared with once daily administered 0.03% Bimatoprost Ophthalmic Solution and once daily administered 0.5% Timolol Ophthalmic Solution concurrently in patients with open-angle glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma or ocular hypertension in one or both eyes
* Eye pressure lowering topical medications are not working
* Visual acuity is at least 0.2 in each eye

Exclusion Criteria:

* Uncontrolled systemic disease
* Any other active eye disease other than glaucoma or ocular hypertension
* Significant visual field loss or evidence of progressive visual field loss within the last year
* Anticipated wearing of contact lenses during the study
* Required chronic use of other ocular medications during the study
* Eye surgery or laser treatment within 12 weeks prior to study enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2010-09-01 (Actual); Study Completion 2010-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Beijing, China

REFERENCES:
- [Background] Ling Z, Zhang M, Hu Y, Yin Z, Xing Y, Fang A, Ye J, Chen X, Liu D, Wang Y, Sun W, Dong Y, Sun X. Safety and efficacy of bimatoprost/timolol fixed combination in Chinese patients with open-angle glaucoma or ocular hypertension. Chin Med J (Engl). 2014;127(5):905-10. PMID 24571886

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.03% Bimatoprost/0.5% Timolol in Same Bottle | 0.03% Bimatoprost and 0.5% Timolol in Separate Bottles
Started | 121 | 114
Completed | 113 | 104
Not Completed | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.03% Bimatoprost/0.5% Timolol in Same Bottle | 0.03% Bimatoprost and 0.5% Timolol in Separate Bottles | Total
Number analyzed (Participants) | 121 | 114 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.73 (14.77) | 44.28 (16.28) | 45.02 (15.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 46 | 92
  Male | 75 | 68 | 143

OUTCOME MEASURES:

1. Primary Outcome: The Difference of Change From Baseline of Mean Diurnal Intraocular Pressure (IOP) Between the Two Treatment Groups at Week 4
Description: The difference of change from baseline of mean diurnal IOP between the 0.03% Bimatoprost/0.5% Timolol in Same Bottle and the 0.03% Bimatoprost and 0.5% Timolol in Separate Bottles at week 4. IOP is a measurement of the fluid pressure inside the eye. Mean diurnal IOP is the average of the IOP values of the study eye (the eye with the highest IOP at baseline) over the 3 time points measured at 8AM, 12PM and 4PM. A negative number change from baseline indicated a reduction (improvement) in IOP. The difference of change from baseline in IOP is presented in the statistical analysis section.
Time Frame: Baseline, Week 4
Population: Intent to Treatment population defined as all patients randomized. One patient in the 0.03% Bimatoprost/0.5% Timolol in Same Bottle group was not included in the analysis.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | 0.03% Bimatoprost/0.5% Timolol in Same Bottle | 0.03% Bimatoprost and 0.5% Timolol in Separate Bottles
Number analyzed (Participants) | 120 | 114
Millimeters of mercury (mmHg)
  Baseline | 25.20 (3.06) | 24.87 (3.88)
  Change from Baseline at Week 4 | -9.38 (4.66) | -8.93 (4.25)
Statistical Analysis 1: Comparison: 0.03% Bimatoprost/0.5% Timolol in Same Bottle vs 0.03% Bimatoprost and 0.5% Timolol in Separate Bottles; A non-inferiority test was performed for comparing the change from baseline in mean diurnal IOP at Week 4 between treatment groups. The null hypothesis was that the mean diurnal IOP change at Week 4 for Group 1 was at least 1.5 mmHg greater than that for Group 2. The hypothesis was tested using a confidence interval approach based on a 2-way analysis of variance (ANOVA) model including factors for treatment and investigator; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of 1.5 mmHg was used. That is, if the upper limit of the 95% confidence interval for the difference in the mean diurnal IOP change between the two groups (Group 1 minus Group 2) is less than 1.5 mm Hg, then the null hypothesis will be rejected. The study had an 85% power; Mean Difference (Final Values) = -0.556, 95% CI 2-sided [-1.68 to 0.57]

ADVERSE EVENTS:
Arm/Group | 0.03% Bimatoprost/0.5% Timolol in Same Bottle | 0.03% Bimatoprost and 0.5% Timolol in Separate Bottles
Serious Adverse Events (participants affected / at risk) | 0/121 | 2/114
Other Adverse Events (participants affected / at risk) | 30/121 | 29/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.03% Bimatoprost/0.5% Timolol in Same Bottle (N=121) | 0.03% Bimatoprost and 0.5% Timolol in Separate Bottles (N=114)
Goitre (Endocrine disorders) | 0 | 1
Ocular hypertension (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.03% Bimatoprost/0.5% Timolol in Same Bottle (N=121) | 0.03% Bimatoprost and 0.5% Timolol in Separate Bottles (N=114)
Conjunctival hyperaemia (Eye disorders) | 26 | 21
Eye pain (Eye disorders) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo